CLINICAL TRIAL: NCT04155866
Title: A Wearable for Post-stroke Rehabilitative Multi-muscle Stimulation Inspired by the Natural Organization of Neuromuscular Control
Brief Title: Comparing the Difference in Muscle Synergies Between Healthy Participants and Chronic Stroke Survivors
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other); City University of Hong Kong (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Cheung Chi Kwan Vincent, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: RIF_Healthy_version 01
Record Dates: First submitted 2019-10-10; First posted 2019-11-07 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy participants: Measurement of lower-limb muscle activation from healthy participants.
  Interventions: Other: Measurement of muscle activation.
- Chronic Stroke Survivors: Measurement of lower-limb muscle activation from chronic stroke survivors
  Interventions: Other: Measurement of muscle activation.

INTERVENTIONS:
Other: Measurement of muscle activation. — Measurement of lower-limb muscle activation during walking for healthy participants.

SUMMARY:
Participants are seeking to unleash the full therapeutic potential of a newly developed, customizable and potentially commericializable 10-channel Functional Electrical Stimulation (FES) to rehabilitate the gait of chronic stroke survivors. Patricipants will utilize the theory of muscle synergies from motor neurosciences, which are defined as neural modules of motor control that coordinate the spatiotemporal activation patterns of multiple muscles, to guide our personal selections of muscles for FES. Before applying FES stimulations to chronic stroke survivors, participants will have to define normal muscle synergies from age-matched healthy control participants (1 session for each participant). After comparing the difference in muscle synergies in both healthy subjects and chronic stroke survivors, participants are attempting to rehabilitate the gait of chronic stroke survivors by using the wearable. Each chronic stroke survivor will undergo 18-session FES training (~ 1 month).

It is hypothesized that FES will promote motor recovery by supplying the missing normal muscle synergies to chronic stroke survivors at their supposed times of activations in each step cycle during interventional training. It is also expected that the walk synergies of the paretic side of chronic stroke survivors should be more similar to healthy muscle synergies at the two post-training time points than before training. The healthy normal muscle synergies will be defined by EMG recordings from the recruited healthy participants.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of long-term adult disability worldwide. The impaired ability to walk post-stroke severely limits mobility and quality of life. Many recently-developed assistive technologies for gait rehabilitation are at present only marginally better at best than traditional therapies in their efficacies. There is an urgent need of novel, clinically viable, and effective gait rehabilitative strategies that can provide even better functional outcome for stroke survivors with diverse presentations.

Among the many new post-stroke interventions, functional electrical stimulation (FES) of muscles remains attractive. FES is a neural-rehabilitative technology that communicates control signals from an external device to the neuromuscular system. There is increasing recognition that rehabilitation paradigms should promote restitution of the patient's muscle coordination towards the normal pattern during training, and FES can achieve this goal when stimulations are applied to the set of muscles whose natural coordination is impaired. For this reason, FES is a very promising interventional strategy. Existing FES paradigms, however, have yielded ambiguous results in previous clinical trials, especially those for chronic survivors, likely because either stimulation were applied only to single or a few muscles, or the stimulation pattern did not mimic the natural muscle coordination pattern during gait. A multi-muscle FES, when applied to a larger functional set of muscles and driven by their natural coordination pattern, can guide muscle activations towards the normal pattern through neuroplasticity, thus restore impairment at the level of muscle-activation deficit.

The aim of our project is to rehabilitate the gait of chronic stroke survivors by delivering stimulations to multiple muscles, in their natural coordination pattern, using our wearable. participants will utilize the theory of muscle synergy from motor neuroscience to guide our personalizable selections of muscles for FES. Muscle synergies are hypothesized neural modules of motor control that coordinate the spatiotemporal activation patterns of multiple muscles. Our customizable FES pattern for each stroke survivor will be constructed based on the normal muscle synergies - identified from age-matched healthy subjects - that are absent in the stroke survivor's muscle pattern during walking. Since muscle synergies represent the natural motor-control units used by the nervous system, reinforcement of their activations through FES should lead to a restoration of normal neuromuscular coordination, thus more natural post-training gait.

ELIGIBILITY:
Inclusion Criteria:

For chronic stroke survivors:

1. Right-handed elderly chronic stroke survivors; age ≥40; ≥6 months post-stroke
2. Unilateral ischemic brain lesions
3. Participants should be able to walk continuously for ≥15 min. with or without assistive aid

For healthy participants:

1. Healthy, right-handed subjects, age ≥40, free from any history of major neurological, musculoskeletal, and psychiatric disorders
2. Able to walk continuously for ≥20 min. without fatigue.

Exclusion Criteria:

For both healthy participants and chronic stroke survivors:

1. Cannot comprehend and follow instructions, or with a score <21 on the mini-mental state exam;
2. Have cardiac pacemaker;
3. Have skin lesions at the locations where FES or EMG electrodes may be attached;
4. Have major depression;
5. Present with severe neglect

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age-matched healthy control subjects will be recruited through advertisements. Chronic Stroke Survivors will be recruited from the local community such as clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Surface electromyographic signals from up to 14 muscles on each side of healthy participants during gait. | The assessment will be performed at 1 week
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.
Surface electromyographic signals from up to 14 muscles on the paretic and non-paretic side during gait. | The assessment will be performed at baseline
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.
Surface electromyographic signals from up to 14 muscles on the paretic and non-paretic side during gait. | The assessment will be performed at 5.5 weeks
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.
Surface electromyographic signals from up to 14 muscles on the paretic and non-paretic side during gait. | The assessment will be performed at 2.5 weeks
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.
Surface electromyographic signals from up to 14 muscles on the paretic and non-paretic side during gait. | The assessment will be performed at 4 weeks
  To assess the muscle synergies, surface EMGs will be recorded from 14 muscles (tibialis anterior (TA), medical gastrocnemius (MG), soleus (SOL), vastus medialis (VM), rectus femoris (RF), hamstrings (HAM), adductor longus (AL), gluteus maximus (GM) lateral gastrocnemius (LG), vastus lateralis (VL), tensor fasciae latae (TFL), erector spinae (ES), external oblique (EO), and latissimus dorsi (LatDor)), using a wireless EMG system (Delsys; 2000 Hz). All electrodes will be securely attached to skin surface using double-sided and medical tapes.

SECONDARY OUTCOMES:
Measuring Gait kinematics from Healthy Participants | The assessment will be performed at 1 week
  Kinematic measurements will be provided by the wearable's IMUs. During assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Measuring Gait kinematics from Chronic Stroke Survivors | The assessment will be performed at baseline
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Measuring Gait kinematics from Chronic Stroke Survivors | The assessment will be performed at 5.5 weeks
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Measuring Gait kinematics from Chronic Stroke Survivors | The assessment will be performed at 2.5 weeks
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Measuring Gait kinematics from Chronic Stroke Survivors | The assessment will be performed at 4 weeks
  During FES sessions, kinematic measurements will be provided by the wearable's IMUs. During sessions of motor-impairment assessments, we will capture more precise kinematics using a 10-camera motion capture system (VICON; 200 Hz). This system tracks the 3D positions of 40 markers placed on the legs and torso, and is equipped with suitable models for reconstructing bilateral angles of the hip, knee and ankle.
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at baseline
  Lower-limb motor function assessment
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at 5.5 weeks
  Lower-limb motor function assessment
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at 2.5 weeks
  Lower-limb motor function assessment
Fugl-Meyer assessment score (lower-limb) | The assessment will be performed at 4 weeks
  Lower-limb motor function assessment
Mini-BEStest | The assessment will be performed at baseline
  Balance test
Mini-BEStest | The assessment will be performed at 5.5 weeks
  Balance test
Mini-BEStest | The assessment will be performed at 2.5 weeks
  Balance test
Mini-BEStest | The assessment will be performed at 4 weeks
  Balance test

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krasovsky T, Levin MF. Review: toward a better understanding of coordination in healthy and poststroke gait. Neurorehabil Neural Repair. 2010 Mar-Apr;24(3):213-24. doi: 10.1177/1545968309348509. Epub 2009 Oct 12. PMID 19822722
- [Background] Peckham PH, Knutson JS. Functional electrical stimulation for neuromuscular applications. Annu Rev Biomed Eng. 2005;7:327-60. doi: 10.1146/annurev.bioeng.6.040803.140103. PMID 16004574
- [Background] Sheffler LR, Chae J. Neuromuscular electrical stimulation in neurorehabilitation. Muscle Nerve. 2007 May;35(5):562-90. doi: 10.1002/mus.20758. PMID 17299744
- [Background] Heller BW, Clarke AJ, Good TR, Healey TJ, Nair S, Pratt EJ, Reeves ML, van der Meulen JM, Barker AT. Automated setup of functional electrical stimulation for drop foot using a novel 64 channel prototype stimulator and electrode array: results from a gait-lab based study. Med Eng Phys. 2013 Jan;35(1):74-81. doi: 10.1016/j.medengphy.2012.03.012. Epub 2012 May 4. PMID 22559959
- [Background] Springer S, Vatine JJ, Wolf A, Laufer Y. The effects of dual-channel functional electrical stimulation on stance phase sagittal kinematics in patients with hemiparesis. J Electromyogr Kinesiol. 2013 Apr;23(2):476-82. doi: 10.1016/j.jelekin.2012.10.017. Epub 2012 Dec 8. PMID 23231828
- [Background] You G, Liang H, Yan T. Functional electrical stimulation early after stroke improves lower limb motor function and ability in activities of daily living. NeuroRehabilitation. 2014;35(3):381-9. doi: 10.3233/NRE-141129. PMID 25227538
- [Background] Zhuang C, Marquez J, Qu H, He X, Lan N (2015) A neuromuscular electrical stimulation strategy based on muscle synergy for stroke rehabilitation. 2015:816-819.
- [Background] Ferrante S, Chia Bejarano N, Ambrosini E, Nardone A, Turcato AM, Monticone M, Ferrigno G, Pedrocchi A. A Personalized Multi-Channel FES Controller Based on Muscle Synergies to Support Gait Rehabilitation after Stroke. Front Neurosci. 2016 Sep 16;10:425. doi: 10.3389/fnins.2016.00425. eCollection 2016. PMID 27695397
- [Background] Barroso FO, Torricelli D, Molina-Rueda F, Alguacil-Diego IM, Cano-de-la-Cuerda R, Santos C, Moreno JC, Miangolarra-Page JC, Pons JL. Combining muscle synergies and biomechanical analysis to assess gait in stroke patients. J Biomech. 2017 Oct 3;63:98-103. doi: 10.1016/j.jbiomech.2017.08.006. Epub 2017 Aug 20. PMID 28882330